CLINICAL TRIAL: NCT00508846
Title: Screening for Gynecologic Cancers Among Women With Hereditary Non-Polyposis Colon Cancer (HNPCC)
Brief Title: Screening for Gynecologic Cancers in Hereditary Nonpolyposis Colorectal Cancer (HNPCC) Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID03-0211
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Colon Cancer
Keywords: Hereditary Non-Polyposis Colon Cancer; Gynecologic Cancers; Genetic Counseling; Questionnaire; Survey; HNPCC
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HNPCC Patients
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Two-part telephone questionnaire lasting about 60 minutes total.
  Other Names: Survey

SUMMARY:
Among women with HNPCC, this study will assess:

1. Knowledge of screening recommendations for endometrial and ovarian cancers.
2. Perceived risk and cancer worries regarding endometrial, ovarian and colorectal cancers.
3. Adherence to screening recommendations for endometrial, ovarian and colon cancers.
4. Perceived benefits,supports and barriers to endometrial and ovarian cancer screening.
5. Patterns of communication about endometrial and ovarian cancer risk within families with HNPCC and with health care providers.
6. Patient preferences for potential cancer screening and cancer prevention strategies related to HNPCC-associated cancers.

DETAILED DESCRIPTION:
Women who are at risk for HNPCC will be recruited to participate in this pilot study.

Women will be invited to participate in the study either through a mailed invitation or during a visit to M.D. Anderson for clinical services or for research purposes.

Women who wish to participate in the study will complete an informed consent, and will subsequently schedule an appointment with a research coordinator to complete the study questionnaire by telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Being female
2. Being 25 years of age or older
3. Having an HNPCC-predisposing mutation and/or having a family history of cancer that meets the Amsterdam or Amsterdam II criteria for HNPCC

Exclusion Criteria:

1. Persons who have tested negative for a known HNPCC-predisposing mutation in their family
2. Persons who have no family HNPCC mutation and have not met the Amsterdam I/II criteria
3. Being younger than 25 years old
4. Note: Women who have had a prior history of colorectal cancer or polyps will not be excluded unless they meet one of the above exclusion criteria.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, age 25 years of age or older, diagnosed with Hereditary Non-Polyposis Colon Cancer (HNPCC).
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2003-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient Responses to Questionnaire | 7 Years
  Outcomes measuring demographics, surveillance behaviors, perceived risk, and cancer worries, screening supports/benefits and barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org